CLINICAL TRIAL: NCT01710917
Title: The Efficacy of Targinact® Treatment With Respect to Quality of Life (Overall Health Assessment) in Chronic Severe Pain Patients Compared to Previous Analgesic Treatment: a Non-interventional, Observational Study.
Brief Title: A Non-interventional, Observational Study for Quality of Life (Overall Health Assessment) in Patients With Chronic Severe Pain During Targinact® Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mundipharma CVA (Other)
Responsible Party: Sponsor
Other Study IDs: OXN9512
Record Dates: First submitted 2012-10-15; First posted 2012-10-19 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Severe Pain
Keywords: Chronic pain; Severe pain; Oxycodon; Naloxon; Opioid-induced constipation; Opioid; Quality of life; Laxative; Analgesic rescue medication
MeSH Terms: conditions — Chronic Pain; Pain; Opioid-Induced Constipation | interventions — oxycodone naloxone combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Targinact® (oxycodon/naloxon)
  Interventions: Drug: Targinact® (oxycodon/naloxon)

INTERVENTIONS:
Drug: Targinact® (oxycodon/naloxon)

SUMMARY:
This non-interventional, observational study evaluates the efficacy of Targinact with regard to quality of life in daily clinical practice in Belgium compared to the previous analgesic treatment.

DETAILED DESCRIPTION:
Patients are treated with Targinact® according to daily clinical practice during at least 12 weeks and are monitored during study 3 visits. Parameters assessed are overall health assessment of the patient, pain relief, constipation, use of laxatives, use of analgesic rescue medication, use of concomitant medication, quality of life and safety of Targinact® treatment. These parameters, except for safety assessment, are compared between Targinact® treatment and previous analgesic treatment.

ELIGIBILITY:
Inclusion criteria:

Patients enrolled in the study are patients who

* are eligible for Targinact® treatment according to the Targinact® SPC AND
* who have previously been treated with WHO step 1, 2 or 3 analgesics

Exclusion criteria are based on the Targinact® SPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary and Secondary care
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-11 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of Targinact® treatment | 12 weeks
  The primary parameter to assess the efficacy of Targinact® treatment with respect to the quality of life (overall health assessment/EQ-VAS) in patients with chronic severe pain compared to previous analgesic treatment is the absolute change in overall health score (0-100) attributed by patients during Targinact® treatment compared to previous analgesic treatment.
  During each visit, patients will be asked to score their overall health state between 0 (worst health state imaginable) and 100 (best health state imaginable). The absolute changes in overall health assessment from baseline at V2 and V3 will be used to compare health assessment during Targinact® treatment.

SECONDARY OUTCOMES:
• To assess pain (NRS) during Targinact® treatment compared to previous analgesic treatment (by physician) | 12 weeks
  To assess pain (NRS) during Targinact® treatment compared to previous analgesic treatment (by physician)
To assess constipation (BFI) during Targinact® treatment compared to previous analgesic treatment (by physician) | 12 weeks
  To assess constipation (BFI) during Targinact® treatment compared to previous analgesic treatment (by physician)
To assess laxative use during Targinact® treatment compared to previous analgesic treatment (by physician) | 12 weeks
  To assess laxative use during Targinact® treatment compared to previous analgesic treatment (by physician)
To assess the use of analgesic rescue medication during Targinact® treatment compared to previous analgesic treatment (by physician) | 12 weeks
  To assess the use of analgesic rescue medication during Targinact® treatment compared to previous analgesic treatment (by physician)
To evaluate the quality of life (EQ-5D questionnaire) during Targinact® treatment compared to previous analgesic treatment (by patient) | 12 weeks
  To evaluate the quality of life (EQ-5D questionnaire) during Targinact® treatment compared to previous analgesic treatment (by patient)
To assess safety of Targinact® treatment (by physician) | 12 weeks
  Safety will be assessed by documentation of adverse events, collected via spontaneous reports and patient documentation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brussels (UZ Brussel), Belgium, Brussels, Belgium

REFERENCES:
- [Derived] Poelaert J, Koopmans-Klein G, Dioh A, Louis F, Gorissen M, Loge D, Van Op den Bosch J, van Megen YJ. Treatment with prolonged-release oxycodone/naloxone improves pain relief and opioid-induced constipation compared with prolonged-release oxycodone in patients with chronic severe pain and laxative-refractory constipation. Clin Ther. 2015 Apr 1;37(4):784-92. doi: 10.1016/j.clinthera.2015.02.010. Epub 2015 Mar 7. PMID 25757607